CLINICAL TRIAL: NCT06331793
Title: Use of a Wearable Device Which Generates an Electromagnetic Pulsed Field for Postoperative Analgesia of Mastectomies
Brief Title: Pulsed Electromagnetic Fields for Analgesia Post Mastectomy
Acronym: Algocare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IEO 1849
Record Dates: First submitted 2024-03-18; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Female Breast Cancer; Post Operative Pain
Keywords: Unilateral mastectomy with reconstruction; Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomization 1:1
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active AlgoCare (Experimental): An active AlgoCare device (that emits a pulsed radio frequency electromagnetic field at 27.1 MHz) will be placed over the surgical dressing using a plaster or bandage for six days.
  Interventions: Device: Active AlgoCare
- Non-active AlgoCare (Placebo Comparator): A non-active AlgoCare device (that doesn't emit pulsed radio frequency electromagnetic field) will be placed over the surgical dressing using a plaster or bandage for six days.
  Interventions: Device: Non-active AlgoCare

INTERVENTIONS:
Device: Active AlgoCare — Device that emits Pulsed Electromagnetic Fields
  Arms: Active AlgoCare
Device: Non-active AlgoCare — Device that doesn't emit Pulsed Electromagnetic Fields
  Arms: Non-active AlgoCare

SUMMARY:
Study aim is to test AlgoCare, a device that uses the technology PEMF (Pulsed ElectroMagnetic Fields) for the treatment of postoperative pain in oncological breast surgery, in order to demonstrate that the use of Algocare in the postoperative period allows for a reduction in pain intensity in terms of Numerical Rating Scale (NRS) score and use of analgesic drugs.

DETAILED DESCRIPTION:
The treatment of postoperative pain is a priority issue for both the doctor and the patient. Obtaining adequate analgesia in the first postoperative days, in fact, is essential for the patient's comfort, but also to promote and accelerate functional recovery and prevent chronic pain, which in the case of breast surgery has a high incidence (20-60 %).

The use of pulsed electromagnetic fields (PEMF) for the treatment of pain and inflammation has been widely studied and validated.

Study aim is to test AlgoCare, a device that uses the technology PEMF (Pulsed ElectroMagnetic Fields), for the treatment of postoperative pain in oncological breast surgery. This is a field of application in which this technique analgesic has never been tested, but in which it could prove valid within a multimodal analgesia protocol, as the pain caused by this type of intervention is predominantly parietal and resulting from tissue trauma caused by the surgical wound. AlgoCare is a non-invasive and non-pharmacological device, developed specifically for treatment of post-operative inflammation and pain, CE certified and registered with the Ministry of Health. It emits a pulsed radio frequency electromagnetic field at 27.1 MHz, a frequency already studied and approved for medical use.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients undergoing unilateral mastectomy with reconstruction and without axillary dissection

Exclusion Criteria:

* Patients with PaceMakers (PMs), Implantable Cardioverter Defibrillators (ICDs), neurostimulators or other active medical devices or metal implants near the application area
* Pregnancy
* Amyloidosis, sarcoidosis, scleroderma, infectious arthritis, Paget's disease or joint tumors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 72 hours
  Difference in mean NRS score between the two arms, at 24 hours and 72 hours after surgery (minimum value: 0, maximum value: 10 - higher scores mean a worse outcome)

SECONDARY OUTCOMES:
Need for analgesic drugs | 3 months
  Compare analgesic drugs use between the two arms
Patient reported pain characteristics | 3 months
  Compare characteristics of pain between the two arms by collection of a questionnaire that describes kind of pain experienced by patient
Number of participants with other symptoms | 3 months
  Compare presence of other symptoms between the two arms by collection of a questionnarie in which patient reports occurence of nausea, vomiting or other symptoms
Need for other drugs | 3 months
  Compare use of drugs (other than analgesic ones) between the two arms
Wound healing timing | 3 months
  Compare days needed to complete wound healing between the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Sances, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy